CLINICAL TRIAL: NCT07333794
Title: Investigating Clients' Understanding and Expectation Reasonableness in Occupational Therapy and Interns' Performance in Health Education and Chief Complaint/Expectation Interviews.
Brief Title: Client Understanding, Expectations, and Intern Performance in Occupational Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202500540B0
Record Dates: First submitted 2025-12-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06

CONDITIONS: Communication
Keywords: Health Education; Interview; Occupational Therapy
MeSH Terms: conditions — Communication; Health Education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psychiatric Clients: Adult psychiatric clients receiving occupational therapy services at the Department of Psychiatry.
  Interventions: Other: Clinical Interview and Occupational Therapy Knowledge (OTK) Health Education Session
- Occupational Therapy Interns: OT students completing clinical internships in psychiatry.
  Interventions: Other: Clinical Interview and Occupational Therapy Knowledge (OTK) Health Education Session
- Clinical Supervisors: Licensed occupational therapists serving as clinical supervisors.
  Interventions: Other: Clinical Interview and Occupational Therapy Knowledge (OTK) Health Education Session

INTERVENTIONS:
Other: Clinical Interview and Occupational Therapy Knowledge (OTK) Health Education Session — This study involves observational procedures, including: (1) a health education session on occupational therapy knowledge (OTK) delivered by occupational therapy interns, and (2) a semi-structured chief complaint and expectation interview conducted with psychiatric clients by interns. Clinical supervisors and external experts evaluate interns' performance using standardized rating scales, which are developed in this study. No therapeutic or experimental interventions are provided to participants.

SUMMARY:
This study aims to investigate psychiatric clients' understanding of occupational therapy (OT), the reasonableness of their expectations regarding OT services, and OT interns' performance in Occupational Therapy Knowledge (OTK) health education and chief complaint/expectation interviews. The project includes developing assessment instruments for client OT knowledge, expectation reasonableness, and intern communication/education performance, followed by data collection in real clinical settings. Clients, clinical supervisors, and external experts will contribute ratings to evaluate instrument validity and reliability. The study will provide foundational evidence for improving OT health education, communication training, and clinical teaching practices.

DETAILED DESCRIPTION:
This study examines (1) psychiatric clients' understanding of occupational therapy (OT), (2) the reasonableness of their expectations toward OT, and (3) OT interns' performance in OTK health education and chief complaint/expectation interviews. The project includes instrument development and clinical data collection in the Department of Psychiatry, Kaohsiung Chang Gung Memorial Hospital.

Substudy 1: Client OT Knowledge and Expectation Reasonableness

Substudy 1 consists of two phases. Phase 1 focuses on developing two tools-the OT Knowledge Assessment and the OT Expectation Reasonableness Scale. A team of clinical OT experts and a psychometrics specialist will identify key domains, generate items, and establish scoring guidelines. Content and face validity will be evaluated by external experts and psychiatric clients.

The OT Knowledge Assessment will measure clients' understanding of OT concepts and service scope. The OT Expectation Reasonableness Scale will assess whether clients' expectations for OT processes and outcomes are clinically appropriate.

Phase 2 collects data from psychiatric clients. OT interns will conduct initial interviews exploring clients' chief complaints and expectations. Clients will complete the OT Knowledge Assessment, and both clinical supervisors and external experts will independently evaluate expectation reasonableness using standardized scoring guidelines. Descriptive statistics will summarize clients' knowledge levels and expectation patterns.

Substudy 2: Intern OTK Health Education and Interview Performance

Substudy 2 includes three phases. Phase 1 develops two performance measures: the OTK Health Education Performance Scale and the Chief Complaint/Expectation Interview Performance Scale. Preliminary domains include communication clarity, individualized education, understanding-checking, information-gathering, clarification, and empathy. Expert review will ensure content and face validity.

Phase 2 evaluates 30 OT interns who will conduct initial interviews with psychiatric clients after receiving standardized training. Clinical supervisors will provide real-time ratings, and external experts will score audio recordings and transcripts. Combined evaluations will provide a more comprehensive assessment of intern performance.

Phase 3 examines reliability of the new scales. Inter-rater reliability (supervisors vs. experts) and intra-rater reliability (experts' repeated scoring) will be assessed using weighted Kappa and intraclass correlation coefficients (ICC).

ELIGIBILITY:
Inclusion Criteria:

1. Occupational Therapy Students: Currently completing a clinical internship in psychiatric occupational therapy.
2. Clinical Supervisors: Willing to participate in the study.
3. Psychiatric Clients:

(1) Age 20 years or older. (2) Diagnosed with a psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition.

(3) Able to understand simple questions and follow three-step commands.

Exclusion Criteria:

1. Occupational Therapy Students: Unwilling to be audio-recorded.
2. Clinical Supervisors: No exclusion criteria.
3. Psychiatric Clients: Unwilling to be audio-recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric clients receiving occupational therapy services in the Department of Psychiatry at Kaohsiung Chang Gung Memorial Hospital.
  Occupational therapy interns completing clinical internships in psychiatric settings.
  Clinical supervisors who observe and evaluate intern performance during clinical interactions.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Occupational Therapy Knowledge Score | Baseline
  Clients' level of understanding of occupational therapy, measured using the Occupational Therapy Knowledge Assessment, which will be developed in this study. Higher scores will indicate greater knowledge of occupational therapy. The score range is not yet finalized.
Occupational Therapy Expectation Reasonableness Score | Baseline
  Clients' expectations regarding occupational therapy processes and outcomes will be evaluated using the Occupational Therapy Expectation Reasonableness Scale, which will be developed in this study. Higher scores will indicate more clinically appropriate expectations. The score range is not yet finalized.
Occupational Therapy Knowledge Health Education Performance Score | Baseline
  Occupational Therapy interns' performance in delivering occupational therapy health education to psychiatric clients will be evaluated using the Occupational Therapy Knowledge Health Education Performance Scale, which will be developed in this study. Higher scores will indicate better performance in delivering health education. The score range is not yet finalized.
Chief Complaint/Expectation Interview Performance Score | Baseline
  Occupational Therapy interns' performance in conducting chief complaint and expectation interviews will be evaluated using the Interview Performance Scale, which will be developed in this study. Higher scores will indicate better interview performance. The score range is not yet finalized.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Hospital, Kaohsiung City, Niaosong Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No